CLINICAL TRIAL: NCT05104697
Title: TMS for Improving Response Inhibition in Adolescents With OCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bradley Hospital (Other)
Collaborators: Butler Hospital (Other); University of Minnesota (Other)
Responsible Party: Principal Investigator, Kristen Benito, Associate Professor (Research), Bradley Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1697181; 5P20GM130452 (NIH)
Record Dates: First submitted 2021-10-09; First posted 2021-11-03 (Actual); Results first posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Investigators will use a within-subject, counterbalanced design comparing TMS vs Sham in a brief 2-visit protocol
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- TMS at visit 1, Sham at visit 2 (Other): At visit 1, participants will receive active TMS using continuous theta burst over the preSMA. At Visit 2, participants will receive sham (fake) TMS in the same location.
  Interventions: Device: Transcranial Magnetic Stimulation
- Sham at visit 1, TMS at visit 2 (Other): At visit 2, participants will receive active TMS using continuous theta burst over the preSMA. At Visit 1, participants will receive sham (fake) TMS in the same location.
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — All teens will receive active TMS; they will be randomly assigned to receive active TMS at either visit 1 or visit 2 (order counterbalanced)

SUMMARY:
The study will examine whether inhibition of the pre-supplementary motor area (pSMA) using transcranial magnetic stimulation (TMS) normalizes activity in pSMA-connected circuits, improves response inhibition, and reduces compulsions in adolescents with OCD.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-18 years
* Presence of OCD, as indicated by score on the Children's Yale-Brown Obsessive-Compulsive Scale
* Patient and one parent speak English fluently (to ensure comprehension of study measures and instructions
* Right-handed
* If taking psychotropic medications, these have been stable for > 6 weeks and are expected to remain stable for the approximately 3-week study protocol
* If currently in psychotherapy, symptom improvement has plateaued (no improvement in the past 6 weeks and symptoms expected to remain stable for the approximately 3-week study protocol)

Exclusion Criteria:

* • Medical conditions contraindicated for TMS or EEG, including history of intracranial pathology, increased intracranial pressure, epilepsy or seizures, traumatic brain injury, brain tumor, stroke, implanted medical devices, possible pregnancy (female of childbearing age not using effective contraception), or any other serious medical condition (note that medical history will be reviewed by a study physician prior to TMS administration)

  * Metal in the head, except mouth (e.g., cochlear implant, implanted brain stimulators, aneurysm clips)
  * Active suicidality or psychosis
  * Existing diagnosis of Bipolar disorder, Autism Spectrum Disorder, mental retardation, or cognitive disability
  * Substance abuse or dependence
  * Taking a stimulant medication (and unwilling to forgo on study visit days)
  * Taking medication with the potential to lower seizure threshold (e.g., neuroleptics, antipsychotics)
  * Patient is a ward of the state
  * Family history of epilepsy
  * History of syncope

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Benito, PhD, Principal Investigator — Bradley Hospital
Locations (1):
- Emma Pendleton Bradley Hospital, Riverside, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a pediatric OCD specialty clinic between March 2022 and March 2023. Note that recruitment began in March 2022 before the first participant was formally enrolled on the study start date of April 1, 2022.
Pre-assignment Details: All enrolled participants were randomly assigned to a study arm.
Period: Overall Study
Arm/Group | TMS at Visit 1, Sham at Visit 2 | Sham at Visit 1, TMS at Visit 2
Started | 3 | 4
Completed | 3 | 3
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Not different from information reported in participant flow
Groups:
- Total: Total of all reporting groups
Arm/Group | TMS at Visit 1, Sham at Visit 2 | Sham at Visit 1, TMS at Visit 2 | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 4 | 7
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.7 (1.2) | 16.3 (1.0) | 15.1 (1.7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 1 | 0 | 1
  Female | 2 | 3 | 5
  Nonbinary | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 7
Children's Yale Brown Obsessive Compulsive Scale (CYBOCS) [Mean (Standard Deviation); unit: units on a scale] — Clinician-rated measure of OCD symptom severity, total score on a 0 to 40 scale, where higher values indicate more severe symptoms.
  units on a scale | 24.0 (1.7) | 24.3 (5.3) | 24.1 (3.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Response Time on Stop Trials of the Stop Signal Task
Description: Computerized task, where shorter response time (in milliseconds) indicates better performance
Time Frame: Change from pre (within 1 hour before) to post (within 1 hour after) intervention
Population: Does not include data from one participant who withdrew prior to completing the measure
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Active TMS: Visits at which participants received active TMS using continuous theta burst over the preSMA. Note that all participants received both Sham and TMS; N for each "group" reflects the entire participant sample.
- Sham (Fake) TMS: Visits at which participants received sham (fake) TMS. Note that all participants received both Sham and TMS; N for each "group" reflects the entire participant sample.
Arm/Group | Active TMS | Sham (Fake) TMS
Number analyzed (Participants) | 6 | 6
milliseconds | -26.2 (102.1) | -31.7 (123.1)

2. Primary Outcome: Change in Frontocentral P3 Amplitude on Electroencephalogram (EEG)
Description: Electroencephalogram (EEG) measured amplitude on successful stop trials of the stop signal task (SST). Calculated by averaging the epochs of successful stop trials time-locked to the stop signal from the midline electrode (Cz).
Time Frame: Change from pre (within 1 hour before) to post (within 1 hour after) intervention
Population: Does not include data from two participants (one withdrew before completing the measure, one could not be analyzed due to error with EEG data capture)
Measure: Mean (Standard Deviation); unit: microvolts (µV)
Arm/Group | Active TMS | Sham (Fake) TMS
Number analyzed (Participants) | 5 | 5
microvolts (µV) | 0.5 (2.9) | 1.5 (2.2)

3. Secondary Outcome: Self-report Symptom Question
Description: Self-rated compulsions on a single-item 0-5 scale, where higher scores indicate more compulsions
Time Frame: post (within 1 hour after) intervention
Population: Does not include one participant who withdrew before completing measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active TMS | Sham (Fake) TMS
Number analyzed (Participants) | 6 | 6
units on a scale | 2.7 (1.4) | 2.5 (2.1)

ADVERSE EVENTS:
Time Frame: Data were collected at one of two study visits that occurred over the course of two weeks
Arm/Group | Active TMS | Sham (Fake) TMS
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active TMS (N=6) | Sham (Fake) TMS (N=6)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Scalp discomfort (Nervous system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This trial has a small sample size; results will need to be confirmed in a larger sample.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-11-19): https://cdn.clinicaltrials.gov/large-docs/97/NCT05104697/Prot_SAP_001.pdf
  • Informed Consent Form (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/97/NCT05104697/ICF_000.pdf